CLINICAL TRIAL: NCT04969263
Title: Immunogenicity of a Third Dose of Either the Moderna COVID-19 Vaccine or Pfizer-BioNTech COVID-19 Vaccine in Kidney Transplant Recipients Who Failed to Respond After Two Previous Doses
Brief Title: COVID-19 Protection After Transplant Pilot Study
Acronym: CPAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAIT COVID19-TB-02; NIAID CRMS ID#: 38865 (Other: DAIT NIAID)
Record Dates: First submitted 2021-07-16; First posted 2021-07-20 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplant Recipients
Keywords: COVID-19 vaccine; SARS-CoV-2 antibody response
MeSH Terms: interventions — BNT162 Vaccine; COVID-19 Vaccines; RNA, Messenger; CVnCoV COVID-19 vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Open label, non-randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BNT162b2 mRNA-based vaccine (Pfizer/BioNTech) (Experimental): The BNT162b2 mRNA-based vaccine was developed to prevent COVID-19, the disease resulting from Severe Acute Respiratory Syndrome coronavirus (SARS-CoV-2) infection. Kidney transplant recipients who had a suboptimal antibody response to the standard two doses of vaccination with Pfizer/BioNTech will receive a third dose of the the same vaccine.
  Administration: One dose administered intramuscularly, upper arm.
  Interventions: Biological: BNT162b2 vaccine (Pfizer/BioNTech)
- mRNA-1273 vaccine (Moderna) (Experimental): The mRNA-1273 vaccine was developed to prevent COVID-19, the disease resulting from Severe Acute Respiratory Syndrome coronavirus (SARS-CoV-2) infection. Kidney transplant recipients who had a suboptimal antibody response to the standard two doses of vaccination with Moderna will receive a third dose of the same vaccine.
  Administration: One dose administered intramuscularly, upper arm.
  Interventions: Biological: mRNA-1273 vaccine (Moderna)

INTERVENTIONS:
Biological: BNT162b2 vaccine (Pfizer/BioNTech) — 30 microgram dose
  Other Names: COMIRNATY (COVID-19 vaccine, mRNA); SARS-CoV-2 mRNA vaccine; Pfizer-BioNTech COVID-19 vaccine
  Arms: BNT162b2 mRNA-based vaccine (Pfizer/BioNTech)
Biological: mRNA-1273 vaccine (Moderna) — 100 microgram dose
  Other Names: SARS-CoV-2 mRNA vaccine; Moderna COVID-19 vaccine; SPIKEVAX (COVID-19 vaccine, mRNA)
  Arms: mRNA-1273 vaccine (Moderna)

SUMMARY:
Antibodies are an important part of the body's defense against infection. Individuals who have no antibodies or very low antibody levels are considered less well protected from Coronavirus Disease 2019 (COVID-19) than those who have higher antibody levels. What level of antibodies is necessary for protection is currently unknown.

Inadequate antibody response to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) vaccination has been described among kidney transplant recipients. The aim of this study is to elicit an antibody response to vaccination against SARS-CoV-2 in kidney transplant recipients who have failed to respond to two doses of either the Moderna COVID-19 vaccine or Pfizer-BioNTech Coronavirus Disease 2019 (COVID-19) vaccine.

DETAILED DESCRIPTION:
This is an open label, non-randomized study in kidney transplant recipients who received two doses of either mRNA COVID-19 vaccine and have a negative (<0.8 U/mL) or low (titer <50 U/mL) SARS-CoV-2 antibody response using the Roche Elecsys® anti-RBD assay. Eligible participants will receive a third dose of the same mRNA vaccine as the prior two doses.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all the following criteria are eligible for enrollment as study participants-

1. Able to understand and provide informed consent;
2. Recipient of kidney transplant ≥12 months prior to enrollment, without treated allograft rejection in the 6 months preceding enrollment;
3. Received 2 doses of either the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine as specified in the respective Food and Drug Administration Emergency Use Authorization (FDA EUAs), >30 days and <8 months prior to enrollment ; and,
4. Negative (antibody titer < 0.8U/mL) or low (antibodies detected at titer ≤ 50 U/mL) response to the vaccine at > 30 days from dose 2 of the Moderna COVID-19 vaccine or the Pfizer BioNTech vaccine, using the Roche Elecsys® anti-Receptor Binding Domain (RBD) assay.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants-

1. Recipient of any number of doses of any COVID vaccine product other than the Moderna COVID-19 vaccine or the Pfizer-BioNTech COVID-19 vaccine;
2. Known history of severe allergic reaction to any component of either the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine;
3. Thrombotic events, myocarditis, or pericarditis temporally associated with prior dose of COVID-19 vaccine;
4. Any change in transplant immunosuppression regimen (drug or dose) in response to suspected or proven rejection within the last 6 months;
5. Significant graft dysfunction;
6. Receipt of any cellular depleting agent (e.g. ATG, Rituximab, Alemtuzumab, Cyclophosphamide) within 12 months preceding enrollment;
7. Receiving systemic immunomodulatory medication(s) for any condition other than transplant;
8. Any untreated active infection, including BK viremia >10^4 copies;
9. Infection with human immunodeficiency virus (HIV);
10. Maintenance immunosuppressive regimen that includes belatacept or abatacept;
11. Recent (within one year) or ongoing treatment for malignancy; or
12. Any past or current medical problems, treatments, or findings which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the candidate's ability to comply with study requirements or may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorry L. Segev, MD, PhD, Study Chair — Department of Surgery, NYU Grossman School of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in: Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: On average, within 24 months after database lock for the trial.
Access Criteria: Open access.
URL: https://www.immport.org/home

REFERENCES:
- [Background] Werbel WA, Boyarsky BJ, Ou MT, Massie AB, Tobian AAR, Garonzik-Wang JM, Segev DL. Safety and Immunogenicity of a Third Dose of SARS-CoV-2 Vaccine in Solid Organ Transplant Recipients: A Case Series. Ann Intern Med. 2021 Sep;174(9):1330-1332. doi: 10.7326/L21-0282. Epub 2021 Jun 15. No abstract available. PMID 34125572
- [Derived] Karaba AH, Morgenlander WR, Johnston TS, Hage C, Pekosz A, Durand CM, Segev DL, Robien MA, Heeger PS, Larsen CP, Blankson JN, Werbel WA, Larman HB, Tobian AAR. Epitope Mapping of SARS-CoV-2 Spike Antibodies in Vaccinated Kidney Transplant Recipients Reveals Poor Spike Coverage Compared to Healthy Controls. J Infect Dis. 2024 May 15;229(5):1366-1371. doi: 10.1093/infdis/jiad534. PMID 38019656
- [Derived] Werbel WA, Karaba AH, Chiang TP, Massie AB, Brown DM, Watson N, Chahoud M, Thompson EA, Johnson AC, Avery RK, Cochran WV, Warren D, Liang T, Fribourg M, Huerta C, Samaha H, Klein SL, Bettinotti MP, Clarke WA, Sitaras I, Rouphael N, Cox AL, Bailey JR, Pekosz A, Tobian AAR, Durand CM, Bridges ND, Larsen CP, Heeger PS, Segev DL; CPAT investigators. Persistent SARS-CoV-2-specific immune defects in kidney transplant recipients following third mRNA vaccine dose. Am J Transplant. 2023 Jun;23(6):744-758. doi: 10.1016/j.ajt.2023.03.014. Epub 2023 Mar 24. PMID 36966905

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Anti-RBD Negative or Low at Study Entry: recipients who have failed to respond to two doses of either the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine.
Period: Overall Study
Arm/Group | All Participants: Anti-RBD Negative or Low at Study Entry
Started | 81
Completed | 72
Not Completed | 9
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 5
Not completed — Physician decision due to both medical and non-medical considerations | 1

BASELINE CHARACTERISTICS:
Groups:
- Anti-RBD Negative or Low at Study Entry: recipients who have failed to respond to two doses of either the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine.
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 49
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 81
Antibody response after 2-dose series of mRNA COVID-19 vaccine [Count of Participants; unit: Participants] — Participants were considered to show negative response after 2-dose series of mRNA COVID-19 vaccine if they had an antibody response <0.8 U/mL at baseline, and low response if ≥0.8 and <50 U/mL. All tests were required to use the Roche Elecsys® anti-RBD assay.
  Participants
    Anti-RBD negative | 39
    Anti-RBD low | 42

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Recipients Who Achieve an Antibody Response >50 U/mL After the Third Dose of mRNA COVID-19 Vaccine
Description: The proportion of participants who achieve an antibody response >50 U/mL after the third dose of vaccine using the Roche Elecsys® anti-RBD assay is considered to show positive response to the intervention, negative response otherwise.
Time Frame: Outcome was measured at 30 days after study intervention (dose 3 vaccination)
Population: All individuals who receive the intervention and have antibody response measured at 30 days after the intervention will be included in the analysis of the primary outcome. For secondary and exploratory outcomes, all individuals who receive the intervention and have that outcome measured will be included.
Measure: Number (95% Confidence Interval); unit: Percentage of participants with response
Groups:
- Anti-RBD Negative or Low at Study Entry: The proportion of recipients who have failed to respond to two doses of either the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine.
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Percentage of participants with response | 69.1 [57.9 to 78.9]

2. Secondary Outcome: Frequency of/Proportion of Participants With Vaccine Reactogenicity (Local or Systemic) and/or Allergy to the mRNA-Based COVID-19 Vaccine
Description: Safety measure status post third dose of mRNA vaccine
Time Frame: Through Day 7 Post-Vaccination (Dose 3)
Measure: Number (95% Confidence Interval); unit: Proportion of participants as percentage
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Proportion of participants as percentage
  Overall Events | 50.6 [39.3 to 61.9]
  Local Reactogenicity | 45.7 [34.6 to 57.1]
  Systemic Reactogenicity | 27.2 [17.9 to 38.2]
  Allergic Reaction | 1.23 [0.03 to 6.69]

3. Secondary Outcome: Frequency of/Proportion of Participants With Any Serious Adverse Events (SAEs) Following the Third Dose of an mRNA Vaccine
Description: Safety measure status post third dose of mRNA vaccine
Time Frame: Through Day 30 Post-Vaccination (Dose 3)
Population: The SAE that occurred through Day 30 post-vaccination (dose 3) was a Urinary Tract Infection that was assessed as unrelated to the study vaccine.
Measure: Number (95% Confidence Interval); unit: Proportion of participants as percentage
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Proportion of participants as percentage | 1.23 [0.03 to 6.69]

4. Secondary Outcome: Proportion of Participants Treated for Acute Cell-Mediated and/or Antibody-Mediated Allograft Rejection (Clinical or Biopsy Proven)
Description: Safety measure status post third dose of mRNA vaccine
Time Frame: Through Day 60 Post-Vaccination (Dose 3)
Measure: Number (97.5% Confidence Interval); unit: Proportion of participants as percentage
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Proportion of participants as percentage | 0 [0 to 4.5]

5. Secondary Outcome: Proportion of Participants Who Develop de Novo Donor-Specific Anti-Human Leukocyte Antigens (HLA) Antibody
Description: Safety measure status post third dose of mRNA vaccine
Time Frame: Through Day 90 Post-Vaccination (Dose 3)
Measure: Number (97.5% Confidence Interval); unit: Proportion of participants as percentage
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Proportion of participants as percentage | 0 [0 to 4.5]

6. Secondary Outcome: Proportion of Participants With Graft Loss
Description: Safety measure status post third dose of mRNA vaccine.
Time Frame: Through Day 60 Post-Vaccination (Dose 3)
Measure: Number (97.5% Confidence Interval); unit: Proportion of participants as percentage
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Proportion of participants as percentage | 0 [0 to 4.5]

7. Secondary Outcome: Occurrence of Death Among Participants
Description: Safety measure status post third dose of mRNA vaccine.
Time Frame: Through Day 60 Post-Vaccination (Dose 3)
Measure: Number (97.5% Confidence Interval); unit: Proportion of participants as percentage
Arm/Group | Anti-RBD Negative or Low at Study Entry
Number analyzed (Participants) | 81
Proportion of participants as percentage | 0 [0 to 4.5]

ADVERSE EVENTS:
Time Frame: AEs are reported for 30 days post vaccine and SAEs for 6 months post vaccine.
Description: Adverse Events temporally associated (24 hours) with the research blood draws and nasopharyngeal swabs will be collected from the time of the screening visit until a participant completes study participation.
  Adverse Events as defined in Section 12.2.1 in the protocol will be collected for 30 days following COVID-19 vaccine administration. Serious Adverse Events will be collected for 6 months following vaccine administration.
  No reported Serious Adverse Events were related to the vaccine.
Groups:
- Anti-RBD Negative or Low at Study Entry: recipients who have failed (negative or low) to respond to two doses of either the Moderna COVID-19 vaccine or Pfizer-BioNTech COVID-19 vaccine.
Arm/Group | Anti-RBD Negative or Low at Study Entry
All-Cause Mortality (participants affected / at risk) | 1/81
Serious Adverse Events (participants affected / at risk) | 12/81
Other Adverse Events (participants affected / at risk) | 57/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-RBD Negative or Low at Study Entry (N=81)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Pyelonephritis (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-RBD Negative or Low at Study Entry (N=81)
Vaccination complication (Injury, poisoning and procedural complications) | 32 (34)
Fatigue (General disorders) | 18 (19)
Headache (Nervous system disorders) | 9 (10)
Lymphocyte count decreased (Investigations) | 9 (9)
Creatinine urine increased (Investigations) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Hyperkaliemia (Metabolism and nutrition disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6)
White blood cell count decreased (Investigations) | 5 (5)
Urinary tract infection (Infections and infestations) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Blood Bicarbonate decreased (Metabolism and nutrition disorders) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 3 (3)
Dizziness (Vascular disorders) | 3 (3)
Injection site erythema (General disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Contusion (Vascular disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/63/NCT04969263/Prot_SAP_001.pdf